CLINICAL TRIAL: NCT06289686
Title: MIRROR Project 44 - Rotator Cuff Repairs With or Without BioEnthesis™ Augmentation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Sparta Biopharma (Unknown); Musculoskeletal Injury Rehabilitation Research for Operational Readiness (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Andrew Sheean, Orthopaedic Surgeon, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2023.080
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Surgery
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BioEnthesis (Experimental): Allogenic, acellular, biphasic allograft (BioEnthesis)
  Interventions: Procedure: Rotator cuff repairs with BioEnthesis augmentation
- Standard of Care (Active Comparator): Standard rotator cuff repair (suture and anchor based technique)
  Interventions: Procedure: Rotator cuff repairs without BioEnthesis augmentation

INTERVENTIONS:
Procedure: Rotator cuff repairs with BioEnthesis augmentation — Rotator cuff repair using BioEnthesis allograft patch
  Arms: BioEnthesis
Procedure: Rotator cuff repairs without BioEnthesis augmentation — Rotator cuff repair using standard of care sutures and anchors
  Arms: Standard of Care

SUMMARY:
Rotator cuff (RC) injuries are particularly prevalent, difficult to repair, and attachment between the bone and tendon is notoriously difficult to achieve. The most common method and current standard of care (SOC) for reattaching connective tissues (e.g., ligaments, tendons) to bone typically involves suture anchor-based techniques, but this is fraught with problems. More specifically, re-tearing of the connective tissue after this procedure occurs in 30-60% of cases, and can be even higher in patients who engage in smoking, have a diagnosis of diabetes, etc. To address these clinical challenges, Sparta Biopharma Inc. (Sparta) developed a unique technology, called BioEnthesis, to improve the connection between the tendon and bone. Pre-clinical in vivo studies demonstrated that the biphasic bovine cancellous matrix regenerated at the bone-soft tissue interface-thereby leading to high structural integrity and will likely lead to reduced re-tear rates over time. The investigators hypothesize that patients in this interventional cohort will experience enhanced mobility, reduced pain, and less re-tears after RC procedures versus a standard suture anchor-based repair.

ELIGIBILITY:
Inclusion Criteria:

* DEERS-eligible
* Adults, between the ages of 18-65 (inclusive)
* Presenting with a rotator cuff tear that is reparable surgically (a reparable tear is defined as tear of the RC where it is possible to bring the retracted tendon edge back to the greater tuberosity of the humerus under minimal tension)
* Ability to undergo surgery to repair rotator cuff tear
* Willingness to commit to study procedures including study intervention and a 12-month follow-up
* Fluency in speaking, reading, comprehending English
* 1-2 tendon full thickness reparable RC tear (full thickness tear is defined as a tear that involves the majority of supraspinatus and less than half of the infraspinatus under minimal tension, with no subscapularis involvement beyond the upper border)

Exclusion Criteria:

* Previous shoulder surgery (excluding acromioplasty or diagnostic arthroscopy)
* Inability to receive an MRI
* Current (within the past 6 months) tobacco user
* Unwilling to remain tobacco free for the duration of the study
* Current lower limb injuries requiring walking assist devices such as crutches and walkers
* Diagnosed with systemic arthritis
* Significant neck pathology
* Active joint or systemic infection
* Currently enrolled, or plans to enroll, in another clinical trial during this study (that would affect the patient's safety or results of this trial)
* Significant muscle paralysis of the shoulder girdle
* Currently pregnant or plans to become pregnant during this study
* Inability of the surgeon to repair the tear with remaining defect no greater than 10 mm in diameter
* Inability of the surgeon to repair the tear with less than 1cm of medialization
* Evidence of other significant shoulder pathology including Type II-IV SLAP lesion, Bankart lesion, Hill Sachs lesion, Grade III osteoarthritis.
* Has a history of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or drug abuse or addiction
* Major medical illness that would preclude undergoing surgery
* Major psychiatric illness or developmental handicap
* Goutallier III classification and above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rates of re-tear | Post-operation at 3-months, 6-months, and 12-months
  Re-tear rates following rotator cuff repair using BioEnthesis versus standard of care. Assessed with (1) 12-month follow-up shoulder MRI and assigning Sugaya Classification, and (2) adverse events evaluation at each follow-up timepoint

SECONDARY OUTCOMES:
Change in the Visual Analogue Scale (VAS) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 3-months, 6-months, and 12-months
  A tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Change in the return to activities of daily living (ADL) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 3-months, 6-months, and 12-months
  A survey asking patients if and when patients have returned to various activities of daily living, such as work, driving, physical/recreational activities.
Change in the Concomitant medications (ConMeds) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 3-months, 6-months, and 12-months
  A survey asking patients to indicate any medications they are taking at the time of the survey (e.g., Acetaminophen, opioids, NSAIDs, etc.)
Change in the Single Assessment Numeric Evaluation (SANE) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 6-months, and 12-months
  The SANE score is a validated patient reported outcome measure. It is a single question score that asks, "how would you rate your condition today as a percentage of normal (0% to 100% scale with 100% being normal)?" The SANE score is collected as standard of care.
Change in the American Shoulder and Elbow Surgeons Standardized Shoulder Form (ASES) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 6-months, and 12-months
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points
Change in the Constant-Murley Score from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 6-months, and 12-months
  The Constant-Murley Score is a multi-item functional scale assessing pain, activities of daily living, range of motion, and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively.
Change in the shoulder immobilization status from before surgery to after surgery | Post-operation at 3-months, 6-months, and 12-months
  A survey asking patients to indicate if they wore a sling after their surgery and for how long they wore their sling.
Change in strength measurements from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 6-months and 12-months
  Strength measurements will be collected using a handheld dynamometer while the arm is in two positions: (1) abduction with the arm in the scapular plane, and (2) external rotation while the arm is adducted and the elbow is flexed to 90 degrees
Change in range of motion measurements from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 6-months and 12-months
  Range of motion measurements will be collected using a goniometer while the arm moves through four movements: (1) forward flexion, (2) abduction, (3) external rotation, and (4) internal rotation
Number of medical events/adverse events after surgery | Day of surgery and post-operation at 3-months, 6-months, and 12-months
  A count of the number of post-operative medical/adverse events for the affected shoulder after the patient's surgery.
Cumulative number of steroid injections after surgery | Post-operation at 3-months, 6-months, and 12-months
  A count of the number of post-operative steroid injections obtained for the affected shoulder after the patient's surgery.
Number of unscheduled visits after surgery | Post-operation at 3-months, 6-months, and 12-months
  A count of the number of clinic visits outside the typical standard of care visits for the affected shoulder after the patient's surgery.
Number of for-cause imaging procedures | Post-operation at 3-months, 6-months, and 12-months
  A count of the number of radiographic imaging obtained, and the type of imaging obtained, for the affected shoulder after the patient's surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dickens, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brooke Army Medical Center, San Antonio, Texas

REFERENCES:
- See also: BioEnthesis Website — https://www.bioenthesis.com/

DOCUMENTS (1):
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT06289686/ICF_000.pdf